CLINICAL TRIAL: NCT02186652
Title: The Effect of Obesity on the Pharmacokinetics of Pantoprazole in Children and Adolescents
Brief Title: PK Study With Pantoprazole in Obese Children and Adolescents
Acronym: PAN01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phillip Brian Smith (Other)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, Phillip Brian Smith, Principal Investigator, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00048765
Record Dates: First submitted 2014-07-03; First posted 2014-07-10 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: obese; children; adolescents; GERD; pharmacokinetic
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity | interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pantoprazole (Other)
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole

SUMMARY:
Multicenter, comparative single-dose pharmacokinetic (PK) study

DETAILED DESCRIPTION:
Evaluate the pharmacokinetics of pantoprazole in obese children and adolescents with gastroesophageal reflux disease (GERD) following administration of an oral dose of pantoprazole.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is between 6 and 17 (inclusive) years of age at the time of consent
2. BMI ≥95th percentile
3. Diagnosis of GERD established prior to 7 days before receipt of study drug dose defined as 1 or more of the following:

   1. clinical symptoms consistent with GERD as determined by the investigator
   2. a diagnosis of erosive esophagitis by endoscopy
   3. esophageal biopsy with histopathology consistent with reflux esophagitis
   4. abnormal pH-metry consistent with reflux esophagitis
   5. other test result consistent with GERD
4. Written informed consent from the parent or legally authorized representative/guardian and participant assent per local IRB recommendation of age-appropriate consent and assent requirements

Exclusion Criteria:

1. Use of pantoprazole, lansoprazole, omeprazole, esomeprazole or rabeprazole within 48 hours prior to dose of study drug
2. Use of fluoxetine, fluvoxamine, ketoconazole, ticlopidine, felbamate, topiramate, valproic acid, phenobarbital, carbamazepine, erythromycin, clarithromycin, grapefruit juice, verapamil, diltiazem, cimetidine, St. John's Wort, rifampin, rifapentine within seven days prior to dose of study drug
3. Consumption of food after midnight on the day of the baseline visit
4. Symptomatic asthma
5. Type I diabetes
6. History of adverse reaction to PPI
7. Impaired hepatic activity as defined as any of the following: AST ≥150 IU/L, ALT ≥150 IU/L, total bilirubin ≥2.0 mg/dl, or alkaline phosphatase ≥600 IU/L
8. Serum creatinine ≥2.0 mg/dL
9. For females of childbearing potential, a positive pregnancy test result
10. Known infection with hepatitis B, C, or HIV
11. Any other condition that, in the opinion of the principal investigator, makes participation unadvised or unsafe.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2014-06-04 (Actual); Primary Completion 2015-09-13 (Actual); Study Completion 2015-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip B Smith, MD, Principal Investigator — Duke Clinical Research Institute
Locations (4):
- United States (4):
  - University of Arkansas, Little Rock, Arkansas
  - Children's Mercy Hospital, Kansas City, Missouri
  - East Carolina University, Greenville, North Carolina
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Shakhnovich V, Smith PB, Guptill JT, James LP, Collier DN, Wu H, Livingston CE, Zhao J, Kearns GL; Best Pharmaceuticals for Children Act - Pediatric Trials Network. Obese Children Require Lower Doses of Pantoprazole Than Nonobese Peers to Achieve Equal Systemic Drug Exposures. J Pediatr. 2018 Feb;193:102-108.e1. doi: 10.1016/j.jpeds.2017.10.011. PMID 29389444

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant for this study began on 8-July-2014. The last participant to complete the study was on 13-September-2015.
Groups:
- Pantoprazole 6-11 Year Old; Pantoprazole 12-17 Year Old: The study design included a screening visit (0-31days prior to baseline), during which informed consent was obtained and blood was collected for isolation of DNA for genotyping.
  During the Baseline Visit (Day 1) included REE measurement (before drug administration using a MedGem indirect calorimeter), study drug administration, and PK evaluation. The MedGem measures oxygen consumption (VO2) to determine resting metabolic rate. Study drug was then administered orally, and repeated blood samples of 1.0 ml each were collected at pre-dose (within 30 minutes), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours (±10 minutes) after dosing. For those participants with the PM CYP2C19 genotype, an additional PK sample was to be obtained at 12 hours after dosing. Between Day 10 and Day 13 after the Baseline Visit, investigators conducted a follow-up call to assess participants' general wellness and to collect Adverse Event (AE) information.
Period: Overall Study
Arm/Group | Pantoprazole 6-11 Year Old | Pantoprazole 12-17 Year Old
Started | 19 | 22
Completed | 17 | 22
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pantoprazole 6-11 Year Old | Pantoprazole 12-17 Year Old | Total
Number analyzed (Participants) | 19 | 22 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 10 (2) | 15 (2) | 12 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 7 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 16 | 19 | 35
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 8 | 12 | 20
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 19 | 22 | 41
Weight [Mean (Standard Deviation); unit: kg] | 60.5 (23.7) | 97.9 (19.6) | 80.6 (28.5)
Weight Percentile [Mean (Standard Deviation); unit: percentile] | 96.8 (3.6) | 97.9 (3.4) | 97.4 (3.5)
Height [Mean (Standard Deviation); unit: cm] | 144.4 (13.9) | 166.6 (7.4) | 156.3 (15.6)
Height Percentile [Mean (Standard Deviation); unit: percentile] | 65.3 (28.9) | 60.9 (29.7) | 62.9 (29.1)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (5.8) | 35.0 (5.0) | 31.7 (6.4)
BMI Percentile [Mean (Standard Deviation); unit: percentile] | 98 (1) | 98 (1) | 98 (1)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Analysis in Obese Children After One Single Oral Dose of Pantoprazole (Cmax).
Description: The pharmacokinetic blood samples will be 1.0 ml each and collected at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, & 8 hours after receiving one dose of Pantoprazole study drug. For those subjects with the poor metabolizer CYP2C19 genotype, an additional PK sample will be obtained at 12 hours after dosing. Here we report Cmax.
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, & 8 hours
Population: All participants with evaluable data.
Measure: Mean (Standard Deviation); unit: mcg/ml
Groups:
- Pantoprazole 6-11 Year Old: same as the participant flow wording.
- Pantoprazole 12-17 Year Old: same as participant flow wording.
Arm/Group | Pantoprazole 6-11 Year Old | Pantoprazole 12-17 Year Old
Number analyzed (Participants) | 18 | 21
mcg/ml | 4.27 (1.43) | 4.1 (1.18)

2. Primary Outcome: Pharmacokinetic Analysis in Obese Children After One Single Oral Dose of Pantoprazole (Tmax).
Description: The pharmacokinetic blood samples will be 1.0 ml each and collected at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, & 8 hours after receiving one dose of Pantoprazole study drug. For those subjects with the poor metabolizer CYP2C19 genotype, an additional PK sample will be obtained at 12 hours after dosing. Here we report Tmax.
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, & 8 hours
Population: All participants with evaluable data.
Measure: Median (Full Range); unit: hours
Arm/Group | Pantoprazole 6-11 Year Old | Pantoprazole 12-17 Year Old
Number analyzed (Participants) | 18 | 21
hours | 2.3 [1.5 to 3] | 2.5 [1.5 to 8]

3. Primary Outcome: PK Sampling
Description: Total number of fresh plasma samples (all participants)
Time Frame: Pre-dose (within 30 minutes), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours (±10 minutes) after dosing
Population: All participants with evaluable data
Measure: Mean (Standard Deviation); unit: Plasma samples
Units Other Than Participants: Plasma samples
Arm/Group | Pantoprazole 6-11 Year Old | Pantoprazole 12-17 Year Old
Number analyzed (Participants) | 19 | 22
Number analyzed (Plasma samples) | 203 | 235
Plasma samples | 11 (2) | 11 (2)

4. Primary Outcome: Drug Concentration in Plasma Samples
Description: Concentration of panto in plasma and concentration of panto sulfone in plasma
Time Frame: Pre-dose (within 30 minutes), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours (±10 minutes) after dosing
Population: All participants with evaluable data
Measure: Mean (Standard Deviation); unit: ng/ml
Units Other Than Participants: plasma samples
Groups:
- Pantoprazole 6-11 Year Old: Edit to include: dosing and any info about the participants experience and how they were treated.
- Pantoprazole 12-17 Year Old: same as other arm description
Arm/Group | Pantoprazole 6-11 Year Old | Pantoprazole 12-17 Year Old
Number analyzed (Participants) | 19 | 22
Number analyzed (plasma samples) | 203 | 235
ng/ml
  Pantoprazole: number analyzed (plasma samples) | 127 | 146
  Pantoprazole | 1558 (1584.6) | 1626.1 (1545.2)
  Pantoprazole Sulfone: number analyzed (plasma samples) | 122 | 134
  Pantoprazole Sulfone | 94.7 (49.1) | 88.7 (36.8)

5. Primary Outcome: Pharmacokinetic Analysis in Obese Children After One Single Oral Dose of Pantoprazole (AUC).
Description: The pharmacokinetic blood samples will be 1.0 ml each and collected at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, & 8 hours after receiving one dose of Pantoprazole study drug. For those subjects with the poor metabolizer CYP2C19 genotype, an additional PK sample will be obtained at 12 hours after dosing. Here we report AUC TBW.
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, & 8 hours
Population: All participants with evaluable data.
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Pantoprazole 6-11 Year Old | Pantoprazole 12-17 Year Old
Number analyzed (Participants) | 18 | 21
mcg*h/mL | 8.87 (4.00) | 11.56 (4.81)

6. Primary Outcome: Pharmacokinetic Analysis in Obese Children After One Single Oral Dose of Pantoprazole (AUC).
Description: The pharmacokinetic blood samples will be 1.0 ml each and collected at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, & 8 hours after receiving one dose of Pantoprazole study drug. For those subjects with the poor metabolizer CYP2C19 genotype, an additional PK sample will be obtained at 12 hours after dosing. Here we report AUC LBW.
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, & 8 hours
Population: All participants with evaluable data.
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Pantoprazole 6-11 Year Old | Pantoprazole 12-17 Year Old
Number analyzed (Participants) | 18 | 21
mcg*h/mL | 5.73 (2.48) | 6.82 (2.70)

7. Primary Outcome: Pharmacokinetic Analysis in Obese Children After One Single Oral Dose of Pantoprazole (CL/F).
Description: The pharmacokinetic blood samples will be 1.0 ml each and collected at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, & 8 hours after receiving one dose of Pantoprazole study drug. For those subjects with the poor metabolizer CYP2C19 genotype, an additional PK sample will be obtained at 12 hours after dosing. Here we report CL/F TBW.
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, & 8 hours
Population: All participants with evaluable data.
Measure: Mean (Standard Deviation); unit: l/h/kg TBW
Arm/Group | Pantoprazole 6-11 Year Old | Pantoprazole 12-17 Year Old
Number analyzed (Participants) | 18 | 21
l/h/kg TBW | 0.14 (0.07) | 0.10 (0.04)

8. Primary Outcome: Pharmacokinetic Analysis in Obese Children After One Single Oral Dose of Pantoprazole (Vd/F).
Description: The pharmacokinetic blood samples will be 1.0 ml each and collected at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, & 8 hours after receiving one dose of Pantoprazole study drug. For those subjects with the poor metabolizer CYP2C19 genotype, an additional PK sample will be obtained at 12 hours after dosing. Here we report Vd/F TBW.
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, & 8 hours
Population: All participants with evaluable data.
Measure: Mean (Standard Deviation); unit: L/kg TBW
Arm/Group | Pantoprazole 6-11 Year Old | Pantoprazole 12-17 Year Old
Number analyzed (Participants) | 18 | 21
L/kg TBW | 0.16 (0.05) | 0.14 (0.04)

9. Primary Outcome: Pharmacokinetic Analysis in Obese Children After One Single Oral Dose of Pantoprazole (Vd/F).
Description: The pharmacokinetic blood samples will be 1.0 ml each and collected at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, & 8 hours after receiving one dose of Pantoprazole study drug. For those subjects with the poor metabolizer CYP2C19 genotype, an additional PK sample will be obtained at 12 hours after dosing. Here we report Vd/F LBW.
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, & 8 hours
Population: All participants with evaluable data.
Measure: Mean (Standard Deviation); unit: L/kg LBW
Arm/Group | Pantoprazole 6-11 Year Old | Pantoprazole 12-17 Year Old
Number analyzed (Participants) | 18 | 21
L/kg LBW | 0.25 (0.09) | 0.25 (0.07)

10. Secondary Outcome: The CYP2C19 Genotype and Its Association With CYP2C19 Phenotype
Description: To examine the association of CYP2C19 genotype and its association with CYP2C19 phenotypes. To characterize the ability of the CYP2C19 genotype to predict pantoprazole plasma clearance, a correlation with CYP2C19 phenotype was explored using both standard linear and nonlinear regression techniques and their respective tests for significance and goodness of fit. In addition, the impact of all covariates on pantoprazole systemic exposure and apparent plasma clearance (e.g., demographic determinants of extent of obesity such as the waist:hip ratio, CYP2C19 genotype, BMI, and REE) was explored using validated population-based PK methods (NONMEM).
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12 hours post-dose
Population: Total analyzed #participants is 38. Total #participants in age groups is 37 excluding one poor-metabolizer.
  Poor metabolizer is defined as a participant who had *2/*2 alleles; intermediate metabolizer is defined as a participant who had *1/*2 or *2/*17 alleles; extensive metabolizer is defined as a participant who had *1/*1 or *1/*17 alleles.
Measure: Median (Full Range); unit: L/h
Groups:
- *2*2 Allele: Poor metabolizer
- *1/*2 Allele: Intermediate Metabolizer
- *1/*1 Allele or *1/*17 Allele: Extensive Metabolizer
Arm/Group | *2*2 Allele | *1/*2 Allele | *1/*1 Allele or *1/*17 Allele
Number analyzed (Participants) | 1 | 16 | 21
L/h | 1.29 [NA to NA] — 1 participant only | 6.00 [2.64 to 11.62] | 8.97 [4.66 to 16.71]

ADVERSE EVENTS:
Time Frame: Adverse events were followed up to 10 days post study dose.
Description: An AE is any untoward medical occurrence in humans, whether or not considered drug-related, which occurs during the conduct of a clinical trial. (Any change in clinical status, ECGs, routine labs, x-rays, physical examinations, etc., that is considered clinically significant by the study investigator is considered an AE.)
Groups:
- 6-11 Year Old Adverse Events; 12-17 Year Old Adverse Events: Study participants were selected from obese children and adolescents ranging in age from 6 17 years (inclusive) and seen in the outpatient clinic for the diagnosis or treatment of GERD. The target enrollment was 40 participants (20 participants 6-11 years of age and up to 20 participants 12 17 years of age). Potential study participants could come from any outpatient clinical setting within participating institutions where children with GERD were seen for evaluation and/or treatment.
Arm/Group | 6-11 Year Old Adverse Events | 12-17 Year Old Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/22
Other Adverse Events (participants affected / at risk) | 1/19 | 6/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6-11 Year Old Adverse Events (N=19) | 12-17 Year Old Adverse Events (N=22)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes